CLINICAL TRIAL: NCT04728841
Title: Clinical Exploration of Clinical Exploration Adeno-associated Virus Vector Expression of Human Coagulation Factor VIII Gene Therapy for Hemophilia A
Brief Title: Gene Therapy for Chinese Hemophilia A
Acronym: HA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2020030
Record Dates: First submitted 2021-01-25; First posted 2021-01-28 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-01

CONDITIONS: Hemophilia A; Gene Therapy
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): Arm of GS001
  Interventions: Genetic: Injection of GS001

INTERVENTIONS:
Genetic: Injection of GS001 — Patients will be enrolled sequentially every 3 weeks or more between cohorts. Dose escalation may occur after a single patient has been safely dosed if the resulting FVIII activity at Week 3 is < 5 IU/dL.The dose levels are as follows:
  1. 2×10^12 vg/kg
  2. 6×10^12vg/kg or other recommended doses
  3. 2×10^13 vg/kg or other recommended doses

SUMMARY:
IHBDH-GTHA-2020 is an open- label, non- randomized study to evaluate the safety, tolerability and kinetics of a single intravenous infusion of GS001 in hemophilia A subjects with <1 IU/dl residual FVIII levels.

DETAILED DESCRIPTION:
IHBDH-GTHA-2020 is a open- label, non- randomized study to evaluate the safety, tolerability and kinetics of GS001 in hemophilia A subjects with residual FVIII levels<1 IU/dl. The first patient will receive a single intravenous infusion of GS001 at a dose level of 2 x 10^12 vg/kg body weight. After three weeks of follow-up for the first patient post infusion of GS001, the dose of GS001 can be adjusted for the other two patients based on the activity level of FVIII:C and safety assessment. Following completion of the first 3 patients received GS001 infusion at 2 x 10^12 vg/kg dose level , the following 3 patients will continue to be enrolled to this dose group if there isn't any unexpected safety risk based on the assessments of FVIII expression and safety profile. The safety data and the activity level of FVIII:C from the first 6 subjects at 2 x 10^12 vg/kg dose level will undergo review by an independent DMC prior to dosing the first subject in the next dose level, DMC may recommend dose escalation to 6 x 10^12 vg/kg body weight or other recommended dose levels.

If the DMC recommends dose escalation to 6 x 10 ^12 vg/kg body weight or other recommended doses, at least 10 weeks of safety data and the activity level of FVIII:C post GS001 infusion from the first 3 subjects in this given dose level will undergo review by an independent DMC prior to dosing the following subjects. Based on the data from the first 3 subjects, DMC may recommend the dose adjustments for subsequent enrolled subjects, and expand the number of subject enrolled. Based on the safety, preliminary efficacy and vector kinetics profile of single intravenous infusions of GS001 at different dose levels in severe hemophilia A patients with endogenous factor FVIII activity levels ≤ 1% in this study, and based on the benefit-risk assessment of the subjects, the dose level to be administered for future larger clinical trial in patients with severe hemophilia A will be determined.

After all enrolled subjects have been followed for at least 12 weeks after intravenous infusion GS001, periodic analysis will be performed. Primary analysis of safety and efficacy will be performed 52 (± 2) weeks after intravenous infusion GS001, and all subjects will receive 52 (± 2) weeks of comprehensive safety and efficacy assessments. After completing the 52 (± 2) week visit (end-of-study visit), subjects will continue to be followed in this study for up to an additional 4 years for long-term safety and efficacy assessment to evaluate the long-term safety and efficacy of GS001 treatment.

A total of 12 to 15 subjects are expected to be enrolled in this study. Subjects will provide informed consent and then undergo screening assessments up to 4-8 weeks prior administration of GS001. All subjects will undergo 260 weeks (5 years) safety observation.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand the purpose and risks of the study and provide informed consent according to national and local privacy laws;
2. Male subjects and ≥ 18 years of age;
3. Have hemophilia A with ≤1 IU/dL (≤1%) endogenous FVIII activity levels at the time of screening. If the screening result is >1% due to previous treatment with FVIII product, then it may be confirmed by documented historical evidence from a certified clinical laboratory demonstrating ≤1% FVIII activity levels ;
4. No history of hypersensitivity or anaphylaxis associated with FVIII product administration;
5. Have no measurable FVII inhibitor as assessed by laboratory two times that were at least one week apart; or documented no prior history of FVIII inhibitor after 150 EDs and no clinical signs or symptoms of decreased response to FVIII infusion ;
6. Have acceptable laboratory values sampled at screening and repeated prior to Day 0; A. Hemoglobin ≥ 11 g/dL; B. Platelets ≥ 100 x 10^9/L; C. AST, ALT, alkaline phosphatase ≤ 1.25 upper limit of normal (ULN); D. Bilirubin ≤ 1.25 ULN; E. Creatinine ≤ 2 mg/dL.
7. Agree to use reliable barrier contraception until the end of the 52 weeks observation period, and three consecutive semen samples are negative for vector sequences after GS001 infusion.

Exclusion Criteria:

1. Have Hepatitis B, hepatitis C or HBsAg, HCVAb, HBV-DNA, HCV-RNA are positive and have clinical significance. Both natural clearers and those who have cleared HCV on antiviral therapy are deemed eligible;
2. Currently Receiving antiviral therapy for hepatitis B and C;
3. Have history of chronic infections or other chronic diseases that may pose a risk to the study participation;
4. Have participated in a previous gene therapy research trial within the last 52 weeks or in a clinical study with an investigational drug within the past 30 days;
5. The subject has any concurrent diseases that cannot tolerate treatments of prednisone or prednisolone as judged by the investigator;
6. History of arterial or venous thromboembolic events (e.g., deep vein thrombosis, non-hemorrhagic stroke, pulmonary embolism, myocardial infarction, arterial embolism);
7. Known inherited or acquired thrombophilia, including conditions associated with increased risk of thromboembolism, such as atrial fibrillation;
8. Major surgery planned in 1 year period following the infusion with GS001;
9. Hypersensitivity to the study vector;
10. Have clinically major diseases or any other unspecified conditions that, in the opinion of the Investigator, makes the subject unsuitable for participating in the study;
11. Patients who are unable or unwilling to comply with the schedule of visits and study assessments described in the clinical protocol;
12. Evidence of other bleeding disorders not associated with hemophilia A.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-03-04 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment- related adverse events | From screening through up to the end of study (about 5 years).
  Number of patients experiencing treatment-related adverse events.
Percentage of subjects in each dose group with newly occurred clinically significant abnormalities in physical examination compared to the baseline. | From the start of study treatment (Day 1) through up to the end of study (about 5 years).
  The number of subjects in each dose group with clinically significant changes in physical examination compared to the baseline.
Changes of Weighted Mean of vital signs (systolic blood pressure [SBP] and diastolic blood pressure [DBP], pulse rate, temperature, respiratory rate) from baseline at each assessment time point for each dose group | From the start of study treatment (Day 1) through up to the end of study (about 5 years).
  The vital signs (SBP, DBP, pulse rate, temperature, respiratory rate) of the subjects were measured. The maximum, minimum, and mean observed values of vital signs (SBP, DBP, pulse rate, temperature, respiratory rate) from the dosing (Day 1) to the end of the study were calculated for each subject.
Changes of Mean Alkaline Phosphatase (ALP), Alanine Amino Transferase (ALT), Aspartate Amio Transferase (AST) from baseline at each assessment time point for each dose group | From the start of study treatment (Day 1) through up to the end of study (about 5 years).
  Blood samples of subjects were collected for the evaluation of liver function throughout this study. All of these parameters are measured to help assess the condition of the liver. For ALP, AST and ALT, the percentage of subjects with the worst post-treatment results in each dose group will be summarized as follows: > 1.0 x ULN ≤ 1.5x ULN; > 1.5 x ULN ≤ 3.0 x ULN; > 3.0 x ULN ≤ 5.0 x ULN; > 5.0 x ULN
Immune response to AAV capsid proteins | From screening period through up to 5 years.
  Changes in the expression levels of neutralizing and binding antibodies of AAV.
Immune response to FVIII transgene | From screening period through up to 5 years.
  The changes of FVIII inhibitor and antibody levels
Viral vector shedding of GS001 | From date of infusion until the date of 3 consecutive documented negative results, assessed up to 1 year.
  The vector shedding in serum, PMBC, saliva, urine, semen and feces will be monitored
Thrombosis risk assessment | From the start of study treatment (Day 1) through up to the end of study (about 5 years).
  For any individual who reaches >150% vector-derived FVIII: C activity levels following the infusion of GS001, laboratory parameters of thrombotic potential will be assessed.

SECONDARY OUTCOMES:
Vector- derived FVIII:C and FVIII antigen levels | From pre-dose phase through up to 1 years post-dose
  Vector- derived FVIII:C and FVIII antigen levels will be measured after dosing.
FVIII usage within 1 year after GS001 infusion | From week 3 to week 52 post GS001 infusion.
  Number of FVIII replacement therapies and total utilization of exogenous FVIII (IU/kg) replacement therapy.
Number of bleeding events requiring exogenous FVIII replacement therapy within 1 year after GS001 infusion | Week 3 to Week 52 post GS001 Infusion
  Number of bleeding events (Spontaneous and Traumatic) requiring exogenous FVIII replacement therapy
Number of bleeding events within 1 year after GS001 infusion | Week 3 to Week 52 post GS001 infusion
  Number of bleeding events (spontaneous or traumatic) including untreated bleeding events

OTHER OUTCOMES:
Long-term FVIII: C activity Level | From year 2 to year 5 post GS001 infusion.
  FVIII: C activity Level at Year 2 (Week 104), Year 3 (Week 156), Year 4 (Week 208), Year 5 (Week 260) post GS001 Infusion
Annualized number of bleeding episodesrequiring exogenous FVIII replacement therapy during long-term follow up. | From year 2 to year 5 post GS001 infusion.
  Annualized number of bleeding episodes requiring exogenous FVIII replacement therapy during every one-year period from Years 2 to Year 5 (week 53 to week 260) post GS001 infusion
Total utilization of FVIII replacement therapy (IU/kg) per year for long-term follow up. | From year 2 to year 5 post GS001 infusion.
  Total utilization of FVIII replacement therapy (IU/kg) per year from Years 2 to Year 5 (week 53 to week 260) post GS001 infusion
Annualized number of bleeding episodes (spontaneous and traumatic) per year for long-term follow up. | From year 2 to year 5 post GS001 infusion.
  Annualized number of bleeding episodes (spontaneous and traumatic) per year including untreated bleeding episodes per year from Years 2 to Year 5 (week 53 to week 260) post GS001 infusion.
Target joints | From date of GS001 infusion until the end of study (about 5 years).
  Number of Target joints, International Hemophilia Prevention and Treatment Collaborative Group (IPSG) MRI score, changes in joint health score changes
Level of Activity and hemophilia activities list | From date of GS001 infusion until the end of study (about 5 years).
  Changes in Level of Activity and hemophilia activities list
Health-related quality of life | From date of GS001 infusion until the end of study (about 5 years).
  Health-related quality of life evaluated by EQ-5D, pain assessment
Health economics evaluation | From date of GS001 infusion until the end of study (about 5 years).
  Health economic parameters include, but are not limited to, the following:number of hospitalizations, number of hospitalization days, number of emergency room visits, number of unscheduled visits, number of days off school or work.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No